CLINICAL TRIAL: NCT04630301
Title: Pleural Manometry for the Characterization of Spontaneous and Tension Pneumothorax
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Medline Industries, Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00256185
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Pneumothorax; Tension Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Measurement of pleural pressure: a. Patients admitted to the Johns Hopkins Hospital with spontaneous, iatrogenic, or tension pneumothorax referred to the Division of Interventional Pulmonology for thoracostomy will be recruited. Using standard sterile technique, a 14fr catheter will be inserted into the pleural space. An electronic manometer (Compass, Medline Industries, Inc.) will be connected in-line to the introducer needle and Ppl will be recorded for 3-5 respiratory cycles. After measurement, the manometer will be removed and the catheter will remain in place per routine standards of practice.

SUMMARY:
Intrapleural pressures have been shown to be a useful clinical predictor in pleural effusions, however it's utility has not been described in pneumothorax. Data on intrapleural pressures in pneumothorax are limited. Furthermore, the pleural pressure in tension pneumothorax is theorized to be greater than atmospheric pressure, though this has never been verified. Pneumothorax is primarily treated with a tube thoracostomy. This observational study will record intrapleural pressures in participants with pneumothorax undergoing a tube thoracostomy. Clinical outcomes of participants will then be monitored for need for pleurodesis, intrabronchial valve placement, and video assisted thoracoscopic surgery (VATS) to identify a correlation with intrapleural pressure.

DETAILED DESCRIPTION:
The rate of hospitalization for spontaneous pneumothorax among people age 14 or older is approximately 227 per million. Spontaneous pneumothorax in the absence of trauma can be further classified as primary spontaneous pneumothorax (PSP) or secondary spontaneous pneumothorax (SSP) based on the absence or presence of underlying structural lung disease, respectively. Though recent studies suggest that in some cases conservative management with close observation is an acceptable treatment, definitive evacuation remains a cornerstone of management for patients who are symptomatic or who have a large pneumothorax. Intrapleural air can be removed by either needle aspiration or introduction of a watersealed catheter into the pleural space. In the event of tension pneumothorax (TP), emergent chest thoracostomy is preferred. In all cases, the goal of treatment remains to re-expand the affected lung, after which the catheter may be removed. If the visceral pleural defect is not healed after 5 days, it is deemed a persistent air leak. In these cases, the chest tube is maintained and more aggressive measures such as pleurodesis, placement of an intrabronchial valve (IBV), or VATS are performed. Unfortunately, there is currently no method to predict which patients will require these more invasive procedures.

The lack of prognostic indicators is not the case in pleural effusions, however. Pleural manometry has been shown to be a useful tool in the management of patients with effusions. Doelken et al. described using an overdamped water manometer or an electronic transducer connected to a thoracentesis catheter for the direct measurement of Ppl with similar accuracy. Traditionally, thoracenteses are aborted after onset of dyspnea or cough, all fluid is drained, or 1 liter of fluid has been removed. This 1 liter limit exists to avoid the feared complicated of reexpansion pulmonary edema. However, monitoring of Ppl during drainage and aborting the procedure once Ppl drops below -20 cmH2O allows for safe drainage of often larger volumes. - Furthermore, it has been demonstrated that Ppl could diagnose non-expandable lung and predict pleurodesis failure in patients with malignant effusion. We recently reported the use of a simple, in-line, digital manometer to measure Ppl in patients with pleural effusion.

Routine use of pleural manometry in the evaluation and management of pneumothorax has not yet been adopted, likely due to the historical difficulty in obtaining measurements and the uncertain clinical benefit pleural manometry provided. It has been found that Ppl in spontaneous pneumothorax was greater in patients that required prolonged drainage. These results were later supported in a study that demonstrated the practicality of measuring Ppl in pneumothorax. Ppl measurements required only up to 30 seconds by using an electronic manometer connected to an intrapleural catheter. Still to date, Ppl in TP have yet to be reported. Ultimately, measurement of Ppl in pneumothorax may help identify patients at increased risk for the need of advanced therapies such as IBV placement, pleurodesis, or VATS. Early identification of these high-risk patients will allow for these interventions to be performed earlier, thus reducing hospital length of stay, associated complications, and health-care costs.

4. Study Procedures

1. Patients admitted to the Johns Hopkins Hospital with spontaneous, iatrogenic, or tension pneumothorax referred to the Division of Interventional Pulmonology for thoracostomy will be recruited. Using standard sterile technique, a 14fr catheter will be inserted into the pleural space. An electronic manometer (Compass, Medline Industries, Inc.) will be connected in-line to the introducer needle and Ppl will be recorded for 3-5 respiratory cycles. After measurement, the manometer will be removed and the catheter will remain in place per routine standards of practice. Outcome data of patients will be collected including duration of chest tube placement, need for pleurodesis, IBV, and referral for VATS. Patient data will be de-identified and stored on the a Johns Hopkins secured (SAFE) desktop. A separate file will also be kept on the SAFE desktop that contains participant Medical Record Numbers to allow for matching of Ppl measurements with clinical outcomes. Once outcome data is collected for a participant, the participant's identifiable information will be removed. A combined waiver of consent and oral consent process will be used. The waiver of consent will allow performance of chest tube placement and the collection of pressure measurements via the manometer without the consent of potential subjects. Subsequently, an oral consent process will be used to invite potential subjects to enroll in the study and to get consent for the use of the pressure data already collected as well as for further data collection from the patients' medical records.
2. No biospecimens will be collected.
3. Patients will be enrolled over the course of 1 year. The study will not impact length of hospitalization.
4. This is a nonblinded study.
5. Patients will continue to receive standard of care treatments. This study may delay catheter placement by mere seconds to accommodate for Ppl measurements, this delay is negligible and
6. will not impact clinical outcomes as even in the case of tension the pleural air will be evacuated via the introducer needle.
7. This study does not include a placebo group.
8. Participant removal criteria include pneumothorax in which Ppl cannot be reliably measured within 30 seconds.
9. Participants removed from the study will continue to receive standard-of-care treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or older admitted to the Johns Hopkins Hospital with clinical or radiographic evidence of new pneumothorax who are referred to Interventional Pulmonology for needle aspiration or tube thoracostomy. TP will be defined as a pneumothorax that results in mean arterial pressure <65 or systolic BP < 90.

Exclusion Criteria:

* bilateral pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or older admitted to the Johns Hopkins Hospital with clinical or radiographic evidence of new pneumothorax who are referred to Interventional Pulmonology for needle aspiration or tube thoracostomy.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Thiboutot, MD, MHS, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Medical School, Ann Arbor, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sahn SA, Heffner JE. Spontaneous pneumothorax. N Engl J Med. 2000 Mar 23;342(12):868-74. doi: 10.1056/NEJM200003233421207. No abstract available. PMID 10727592
- [Background] MacDuff A, Arnold A, Harvey J; BTS Pleural Disease Guideline Group. Management of spontaneous pneumothorax: British Thoracic Society Pleural Disease Guideline 2010. Thorax. 2010 Aug;65 Suppl 2:ii18-31. doi: 10.1136/thx.2010.136986. No abstract available. PMID 20696690
- [Background] Bobbio A, Dechartres A, Bouam S, Damotte D, Rabbat A, Regnard JF, Roche N, Alifano M. Epidemiology of spontaneous pneumothorax: gender-related differences. Thorax. 2015 Jul;70(7):653-8. doi: 10.1136/thoraxjnl-2014-206577. Epub 2015 Apr 27. PMID 25918121
- [Background] Brown SGA, Ball EL, Perrin K, Asha SE, Braithwaite I, Egerton-Warburton D, Jones PG, Keijzers G, Kinnear FB, Kwan BCH, Lam KV, Lee YCG, Nowitz M, Read CA, Simpson G, Smith JA, Summers QA, Weatherall M, Beasley R; PSP Investigators. Conservative versus Interventional Treatment for Spontaneous Pneumothorax. N Engl J Med. 2020 Jan 30;382(5):405-415. doi: 10.1056/NEJMoa1910775. PMID 31995686
- [Background] Doelken P, Huggins JT, Pastis NJ, Sahn SA. Pleural manometry: technique and clinical implications. Chest. 2004 Dec;126(6):1764-9. doi: 10.1378/chest.126.6.1764. PMID 15596671
- [Background] Feller-Kopman D, Berkowitz D, Boiselle P, Ernst A. Large-volume thoracentesis and the risk of reexpansion pulmonary edema. Ann Thorac Surg. 2007 Nov;84(5):1656-61. doi: 10.1016/j.athoracsur.2007.06.038. PMID 17954079
- [Background] Light RW, Jenkinson SG, Minh VD, George RB. Observations on pleural fluid pressures as fluid is withdrawn during thoracentesis. Am Rev Respir Dis. 1980 May;121(5):799-804. doi: 10.1164/arrd.1980.121.5.799. PMID 7406313
- [Background] Lan RS, Lo SK, Chuang ML, Yang CT, Tsao TC, Lee CH. Elastance of the pleural space: a predictor for the outcome of pleurodesis in patients with malignant pleural effusion. Ann Intern Med. 1997 May 15;126(10):768-74. doi: 10.7326/0003-4819-126-10-199705150-00003. PMID 9148649
- [Background] Lee HJ, Yarmus L, Kidd D, Amador RO, Akulian J, Gilbert C, Hughes A, Thompson RE, Arias S, Feller-Kopman D. Comparison of pleural pressure measuring instruments. Chest. 2014 Oct;146(4):1007-1012. doi: 10.1378/chest.13-3004. PMID 24853674
- [Background] Herrejon A, Inchaurraga I, Vivas C, Custardoy J, Marin J. Initial pleural pressure measurement in spontaneous pneumothorax. Lung. 2000;178(5):309-16. doi: 10.1007/s004080000034. PMID 11147314
- [Background] Kaneda H, Nakano T, Murakawa T. Measurement of intrapleural pressure in patients with spontaneous pneumothorax: a pilot study. BMC Pulm Med. 2019 Dec 30;19(1):267. doi: 10.1186/s12890-019-1038-9. PMID 31888739
- [Derived] Latifi A, Wang D, Backer ED, Madisi N, Chopra A, Kapp CM, Wayne M, Howe J, Pai C, Yarmus L, Feller-Kopman D, Thiboutot J. Pleural Manometry in Pneumothorax: Evaluating Tension Physiology and Predicting Outcomes. Chest. 2025 Oct 10:S0012-3692(25)05492-3. doi: 10.1016/j.chest.2025.09.121. Online ahead of print. PMID 41076067

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Measurement of Pleural Pressure
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Measurement of Pleural Pressure
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pleural Pressure (Ppl) Prior to Evacuation of Pleural Air
Description: Ppl is reported in centimeters of water (cmH2O). The normal pleural pressure (Ppl), the pressure within the space between the lung and chest wall, is typically subatmospheric, ranging from -3 to -5 cmH2O. This negative pressure is crucial for keeping the lungs inflated and facilitating normal breathing. In this study, all subjects have pneumothorax so will have abnormal Ppl greater than -3. Tension pneumothorax will have a positive Ppl. There is no known 'normal' or 'expected' value.
Time Frame: Upon needle insertion into the pleural space and for 5 breath cycles, up to 60 seconds
Measure: Mean (Standard Deviation); unit: cmH2O
Groups:
- Tension Participants: Tension group of pneumothorax subjects
- Non-tension Participants: Non-Tension group of pneumothorax subjects
Arm/Group | Tension Participants | Non-tension Participants
Number analyzed (Participants) | 9 | 28
cmH2O | 7.44 (6.37) | -1.79 (4.49)

2. Secondary Outcome: Duration (Days) of Chest Tube Placement
Description: Number of days that chest tube is in place.
Time Frame: Up to 30 days
Population: Participants with data collected
Measure: Mean (Full Range); unit: days
Arm/Group | Measurement of Pleural Pressure
Number analyzed (Participants) | 33
days | 4.30303 [0 to 27]

3. Secondary Outcome: Referral for Pleurodesis
Description: Was the patient referred for pleurodesis (yes/no). Outcome value is for "yes" responses.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tension Participants | Non-tension Participants
Number analyzed (Participants) | 9 | 28
Participants | 1 | 4

4. Secondary Outcome: Intrabronchial Valve (IBV) Placement
Description: Was the patient treated with an intrabronchial valve (yes/no). Outcome value is for "yes" responses.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Measurement of Pleural Pressure
Number analyzed (Participants) | 37
Participants | 3

5. Secondary Outcome: Referral for Video Assisted Thoracoscopic Surgery (VATS)
Description: Was the patient referred for video assisted thoracoscopic surgery (yes/no). Outcome value is for "yes" responses.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Measurement of Pleural Pressure
Number analyzed (Participants) | 37
Participants | 1

ADVERSE EVENTS:
Time Frame: Up to 30 days
Arm/Group | Measurement of Pleural Pressure
All-Cause Mortality (participants affected / at risk) | 6/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT04630301/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT04630301/ICF_001.pdf